CLINICAL TRIAL: NCT00127998
Title: Characterization of Novel Molecular Tools for the Epidemiological Surveillance of Antimalarial Drug Resistance in Mali
Brief Title: Antimalarial Drug Resistance in Mali
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Malaria Research and Training Center, Bamako, Mali (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDC-NCID-4314
Record Dates: First submitted 2005-07-07; First posted 2005-08-09 (Estimated); Last update posted 2006-08-16 (Estimated); Status verified 2006-08

CONDITIONS: Malaria
Keywords: malaria; Plasmodium falciparum; drug resistance; antimalarials; genotype; treatment outcome
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Chloroquine; fanasil, pyrimethamine drug combination; Amodiaquine; amodiaquine, artesunate drug combination; sulfadoxine-pyrimethamine-artesunate; Artemether, Lumefantrine Drug Combination; Mefloquine

INTERVENTIONS:
Drug: chloroquine
Drug: sulfadoxine-pyrimethamine
Drug: amodiaquine
Drug: amodiaquine+artesunate
Drug: amodiaquine+sulfadoxine-pyrimethamine
Drug: sulfadoxine-pyrimethamine+artesunate
Drug: artemether-lumefantrine
Drug: mefloquine

SUMMARY:
Resistance of Plasmodium falciparum (malaria) to current antimalarial drugs and the continuing development of resistance to new antimalarial formulations is one of the major obstacles to effective malaria control and case management. Efficient, comprehensive and validated methods for monitoring drug resistance in advance of the development of resistance to the antimalarial drugs that are in use are urgently needed. Molecular markers of genetic polymorphisms that give rise to resistant P. falciparum parasites and methods in population genetics for evaluating the data can be valuable tools for monitoring drug resistance in the field. This study aims to:

1. Prospectively measure the in vivo response of P. falciparum malaria in Mali to several different antimalarial drugs and drug combinations: chloroquine (CQ), sulfadoxine-pyrimethamine (SP), amodiaquine (AQ), sulfadoxine-pyrimethamine in combination with amodiaquine (SP/AQ), amodiaquine in combination with artesunate (AQ/AS), sulfadoxine-pyrimethamine in combination with artesunate (SP/AS), and artemether-lumefantrine (Co-artem). In one site with preliminary data showing a high rate of P. falciparum resistance to mefloquine (MQ), this drug will also be tested.
2. Measure the frequencies of molecular markers for antimalarial drug resistance, and examine how those results relate to the efficacy of these drugs in treating clinical malaria
3. Measure drug levels at 3 days and correlate with efficacy results.
4. Examine early clinical, parasitologic, and clinical predictors of late treatment failure.
5. Use the knowledge gained in Aims 1-3 to develop a molecular tool for a countrywide resistance surveillance system for antimalarial drugs.

DETAILED DESCRIPTION:
Resistance of Plasmodium falciparum to current antimalarial drugs and the continuing development of resistance to new antimalarial formulations is one of the major obstacles to effective malaria control and case management. Parasite populations are highly resistant to chloroquine on an almost worldwide basis (Central America and Haiti being the exceptions) and resistance to the next line of treatment, SP, is widespread in Asia and large parts of East Africa and South America. SP is also now recommended for use as intermittent preventative treatment (IPT) in pregnancy, which adds to concerns about the development and spread of SP resistance. More expensive combination drug therapy using artesunate and other antimalarials in combination is increasingly being recommended in an effort to extend the useful life of drugs and to slow the spread of antimalarial drug resistance. In all likelihood, resistance will eventually emerge for any new single drug or combination formulation that we deploy in the field.

Given the above, efficient, comprehensive and validated methods for monitoring drug resistance in advance of the development of resistance to the antimalarial drugs that are in use are urgently needed. Such methods would help malaria control and prevention programs in guiding national treatment recommendations and policies. Integrating laboratory expertise, analytic methods based on population genetics, and more traditional methods of surveillance for anti-malarial drug resistance (e.g. in vivo drug efficacy studies) and networking with national and international partners will result in a multidisciplinary, geographically diverse team approach to assessing and monitoring drug resistant malaria, as well as developing and validating molecular methods. This type of effort will greatly assist in maximizing the useful life span of antimalarial drugs and in providing evidence-based guidance for drug policy decisions.

Specific Aims:

1. Prospectively measure the in vivo response of P. falciparum malaria in Mali to CQ, SP, AQ, SP/AQ in combination, AQ/artesunate (AS) in combination, SP/AS, and artemether-lumefantrine (Co-artem). In one site with preliminary data showing a high rate of P. falciparum resistance to MQ, MQ will also be tested.
2. Measure the frequencies of dihydrofolate reductase (dhfr), dihydropteroate synthetase (dhps), P. falciparum chloroquine resistance transporter (pfcrt) and P. falciparum multi-drug resistant (pfmdr 1) genotypes and establish their relationship with in vivo resistance to SP (dhfr and dhps), CQ, AQ, SP/AQ, AQ/AS, SP/AS, and MQ.
3. Measure drug levels at 3 days and correlate with in vivo efficacy results.
4. Examine early clinical, parasitologic, and clinical predictors of late treatment failure.
5. Use the knowledge gained in Aims 1-3 to develop a molecular tool for a countrywide resistance surveillance system for SP, AQ, and MQ.

Study Design:

The study will entail two consecutive years of prospective 28 day in vivo drug efficacy studies carried out during the rainy season in three different malaria transmission sites: Koro (rural town with 71% of resistance to MQ at a lower dose of 15 mg/kg), Pongono (rural town with little exposure to antimalarials) and Faladje (rural village with > 30% of chloroquine resistance). Children aged 6-59 months with clinical symptoms consistent with malaria will be enrolled in the study after screening for fever (axillary temperature >=37.5 C) and malaria asexual parasites identified by microscopic examination of thick blood films.

Blood spotted onto filter papers will be collected prior to treatment and during follow up. These filter paper samples will be used for the molecular detection of drug resistance-conferring gene polymorphisms as well as the HPLC detection and quantification of the respective drugs and their relevant metabolites. In vivo data interpretation will be done using the WHO 28-day protocol (WHO, 2003) and molecular markers will be used for the determination of the genotype resistance index (GRI). Venous blood will be collected at enrollment and at the time of in vivo failure to measure in vitro drug efficacy and cryopreserve parasites to search for novel molecular markers to new antimalarial drugs.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6-59 months
* Absence of severe malnutrition (defined as a child whose weight-for-height is below 3 standard deviations of less than 70% of the median of World Health Organization (WHO) reference values, or who has symmetrical edema involving at least the feet)
* A slide-confirmed infection with P. falciparum only (i.e. no mixed infections)
* Initial parasite density between 2,000 and 200,000 asexual parasites per microliter.
* Absence of general danger signs among children < 5 years (inability to drink or breastfeed; vomiting everything; recent history of convulsions; lethargy or unconsciousness; inability to sit or stand up) or other signs of severe and complicated falciparum malaria according to WHO definitions
* Measured axillary temperature ≥ 37.5 °C
* Ability to attend stipulated follow-up visits
* Informed consent provided by parent/guardian
* Absence of history of hypersensitivity reactions to any of the drugs being evaluated

Exclusion Criteria:

* Aged < 6 or >59 months
* Severe malnutrition (defined as a child whose weight-for-height is below 3 standard deviations of less than 70% of the median of WHO reference values, or who has symmetrical edema involving at least the feet)
* No slide confirmed infection with P. falciparum or a mixed infection that includes a non P. falciparum species
* Initial parasite density < 2,000 or > 200,000 asexual parasites per microliter.
* Presence of general danger signs among children < 5 years (inability to drink or breastfeed; vomiting everything; recent history of convulsions; lethargy or unconsciousness; inability to sit or stand up) or other signs of severe and complicated falciparum malaria according to WHO definitions
* Measured axillary temperature <37.5 °C
* Inability to attend stipulated follow-up visits
* Unwilling to provide informed consent provided by parent/guardian
* History of hypersensitivity reactions to any of the drugs being evaluated

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1011
Dates: Start 2005-07

PRIMARY OUTCOMES:
Early Treatment Failure (ETF, defined as: Development of danger signs or severe malaria on Day 1, 2, or 3, in the presence of parasitemia
Parasitemia on Day 2 higher than Day 0 count irrespective of axillary temperature
Parasitemia on Day 3 with axillary temperature ≥37.5°C
Parasitemia on Day 3 ≥ 25% of count on Day 0
Late Clinical Failure (LCF), defined as: Development of danger signs or severe malaria from Day 4 to Day 28 in the presence of parasitemia, without previously meeting any of the criteria of ETF
Presence of parasitemia and axillary temperature ≥37.5° C on any day from Day 4 to Day 28, without previously meeting any of the criteria of ETF
Late parasitological failure (LPF), defined as: Presence of parasitemia on Day 14 to Day 28 and axillary temperature <37.5°C without previously meeting any of the criteria of ETF or LCF
Adequate Clinical and Parasitological Response (ACPR), defined as: Absence of parasitemia on Day 28 irrespective of axillary temperature, without previously meeting any of the criteria of ETF, LCF or LPF

SECONDARY OUTCOMES:
Frequencies of dhfr, dhps, pfcrt and pfmdr1 P. falciparum genotypes and relationship with in vivo resistance to SP (dhfr and dhps), CQ, AQ, SP/AQ, AQ/AS, SP/AS, and MQ
Drug levels at 3 days and correlation with in vivo efficacy results

CONTACTS AND LOCATIONS:
Overall Officials: Robert D. Newman, MD, MPH, Principal Investigator — Centers for Disease Control and Prevention; Kassoum Kayentao, MD, MSPH, Principal Investigator — Malaria Research and Training Center, Bamako, Mali; John Barnwell, PhD, MPH, Principal Investigator — Centers for Disease Control and Prevention; Ogobara Doumbo, MD, PhD, Principal Investigator — Malaria Research and Training Center, Bamako, Mali
Locations (3):
- Mali (3):
  - Faladje Missionary Dispensary, Faladié
  - Koro Health Center, Koro
  - Pongono Community Health Center, Pongono

REFERENCES:
- [Background] WHO. Assessment and Monitoring of Antimalarial Drug Efficacy for the Treatment of Uncomplicated Falciparum Malaria. Geneva: World Health Organization, 2003
- [Background] Plowe CV. Monitoring antimalarial drug resistance: making the most of the tools at hand. J Exp Biol. 2003 Nov;206(Pt 21):3745-52. doi: 10.1242/jeb.00658. PMID 14506209
- [Background] Wernsdorfer WH, Noedl H. Molecular markers for drug resistance in malaria: use in treatment, diagnosis and epidemiology. Curr Opin Infect Dis. 2003 Dec;16(6):553-8. doi: 10.1097/00001432-200312000-00007. PMID 14624105
- [Background] Djimde A, Doumbo OK, Steketee RW, Plowe CV. Application of a molecular marker for surveillance of chloroquine-resistant falciparum malaria. Lancet. 2001 Sep 15;358(9285):890-1. doi: 10.1016/S0140-6736(01)06040-8. No abstract available. PMID 11567708
- [Background] Djimde A, Doumbo OK, Cortese JF, Kayentao K, Doumbo S, Diourte Y, Coulibaly D, Dicko A, Su XZ, Nomura T, Fidock DA, Wellems TE, Plowe CV. A molecular marker for chloroquine-resistant falciparum malaria. N Engl J Med. 2001 Jan 25;344(4):257-63. doi: 10.1056/NEJM200101253440403. PMID 11172152